CLINICAL TRIAL: NCT05430178
Title: Understanding the Metabolic Pathology of Pediatric Obesity and NAFLD
Brief Title: Metabolic Pathology of Pediatric NAFLD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oklahoma (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 14018; 1R01DK129656-01A1 (NIH)
Record Dates: First submitted 2022-06-01; First posted 2022-06-24 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Nonalcoholic Fatty Liver; Nonalcoholic Steatohepatitis; Obesity
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Obesity

STUDY DESIGN:
Intervention Model Description: Cross-sectional design in which all participants receive all interventions in the form of short-term observations following oral consumption of test materials.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- NAFLD (Experimental): Participants in the pediatric NAFLD clinic
  Interventions: Other: Oral sugar tolerance test; Other: De novo lipogenesis test; Other: Gluconeogenesis test
- Ob control (Experimental): Participants with obesity, without NAFLD
  Interventions: Other: Oral sugar tolerance test; Other: De novo lipogenesis test; Other: Gluconeogenesis test
- NW control (Experimental): Participants in the normal range for body weight, without NAFLD
  Interventions: Other: Oral sugar tolerance test; Other: De novo lipogenesis test; Other: Gluconeogenesis test
- Liver control (Experimental): Participants undergoing liver biopsy or liver surgery, without NAFLD
  Interventions: Other: Oral sugar tolerance test; Other: De novo lipogenesis test; Other: Gluconeogenesis test

INTERVENTIONS:
Other: Oral sugar tolerance test — Measurement of glucose and insulin for calculation of insulin sensitivity
Other: De novo lipogenesis test — Oral consumption of deuterated water to measure incorporation of label into lipids
Other: Gluconeogenesis test — Oral consumption of 13C-labeled glycerol to measure incorporation into glucose

SUMMARY:
Nonalcoholic fatty liver disease (NAFLD) is now the most common liver disease worldwide and affects nearly 40% of obese youth and up to 10% of the general pediatric population. Some features of NAFLD are similar in children and adults, yet fibrosis and inflammation are more common in the portal zone and occur earlier in pediatric NAFLD patients than adults. This portends a rapid progression to end-stage liver disease in early adulthood. For the majority of children with NAFLD, mechanisms driving the origin and rapid progression of disease remain unknown. Thus, there is a critical, unmet need to study the specific underlying patterns of metabolic and molecular changes in the liver underlying the development and progression unique to children with NAFLD.

This proposal will test the hypotheses that children with NAFLD have excess glucose and lipid produced by the liver, that those events are regulated by specific variations in the amount and location of RNAs and proteins in liver, and that the concentration of specific micro-RNAs in the blood can be used as a biomarker for NAFLD in pediatric patients.

DETAILED DESCRIPTION:
This project uses a cross-sectional design with a single testing period without a formal intervention (e.g., diet, drug, exercise) or natural follow-up period. Participants with nonalcoholic fatty liver disease (NAFLD), and age-matched control groups classified as either obese (Ob control) or normal weight (NW control) will complete all metabolic and descriptive tests, including blood analyses.

The NAFLD group will also have a liver biopsy as part of their standard clinical care; a portion of the biopsy will be used for the research testing. The Ob and NW control groups will not undergo liver biopsy. To provide a set of reference liver samples to compare with the NAFLD group, we will enroll a "liver control" group, consisting of age-matched patients who are scheduled to have a cholecystectomy with liver biopsy or are undergoing liver resection for tumor removal.

ELIGIBILITY:
Inclusion Criteria:

* Age: All participants must be 10.0 to 20.9 years old at the time of enrollment.
* Sex: Male and Female participants are eligible.
* Race/Ethnicity: Participants of all racial/ethnic identities will be recruited.
* Body mass index (BMI): Participants must be either in the normal weight (NW control group) or obese [Ob control, nonalcoholic fatty liver disease (NALFD) groups] range for BMI percentile. BMI percentile will be calculated from age- and sex-specific growth charts for children.
* NAFLD status: The NAFLD group participants will be eligible if they are scheduled for liver biopsy for clinical reasons and their histopathology report confirms a diagnosis of NAFLD. NW control, and Ob control, and Liver control participants must not have diagnosed NAFLD.

Exclusion Criteria:

* Chronic illness: Participants will not be able to participate if they have conditions that are likely to affect metabolic variables (either directly or due to required medications) or result in them being unable to complete the required tests. Such conditions could include, but are not limited to, untreated hypothyroidism or other endocrine disorders, rheumatoid arthritis requiring steroids or limiting mobility, cardiovascular disease, stroke, or cardiac failure, neurological disorders such as multiple sclerosis, cancer, liver diseases other than NAFLD (e.g., Wilson's disease), other organ disorders, or orthopedic conditions that limit physical activity.
* Acute illness: Participants will not be able to participate if they develop acute conditions that are likely to affect metabolic outcomes (either directly or due to required medications) or result in them being unable to participate; e.g., respiratory illness, infectious disease, fever, accident resulting in bone fractures, myocardial infarction, major depression. If such conditions resolve and there are no longer risks or likelihood of adverse effect on the study outcomes, participants may be rescheduled for testing.
* Medications and nutritional supplements: Medications, vitamins, or supplements that have known effects on the primary outcomes will be cause for exclusion. Examples include weight loss medications, glucocorticoids, or experimental medications used to correct a metabolic or hepatic condition. Medications used to control asthma, allergies, anxiety, depression, attention deficit disorder, menstrual cycle, hypothyroidism, gastric reflux, hypertension, and sleep will be allowed. Participants who are taking medications for treatment of acute illness or conditions such as cold, flu, injury, or infection will be rescheduled after they complete their treatment course.
* Pregnancy: Evidence of pregnancy or intent to become pregnant during the study is cause for exclusion.
* Smoking, alcohol abuse, or illicit drug abuse: Participants who smoke or have signs or symptoms of alcohol or substance abuse will be excluded.

Ages: 10 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-05-25 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
De novo lipogenesis | Day 1
  Measurement of the rate of newly synthesized triglycerides in plasma using deuterated water
Gluconeogenesis | Day 1
  Measurement of the rate newly synthesized glucose in circulation using labeled glycerol and deuterated water
Serum microRNA | Day 1
  Abundance of microRNAs in serum using a broad profiling platform and real-time quantitative polymerase chain reaction tests for confirming individual miRNAs
Abundance of liver collagen | Day 1
  Abundance of collagen in liver biopsy sections, using Second Harmonic Generation microscopy
Liver mitochondrial flux | Day 1
  Reported as the fluorescent lifetime redox ratio (FLIRR), which is calculated from measurements of free and bound NADH and FAD in liver biopsy sections, using fluorescence lifetime imaging microscopy
Insulin sensitivity | Day 1
  Calculated value of insulin sensitivity, using the oral minimal model and serial concentrations of glucose and insulin during an oral sugar tolerance test

SECONDARY OUTCOMES:
Targets of microRNA-122 | Day 1
  Transcripts bound to microRNA-122, measured using high-throughput sequencing of cross- linked immunoprecipitates (HITS-CLIP)
Liver transcriptomics | Day 1
  Spatial distribution of messenger RNAs in liver biopsies

OTHER OUTCOMES:
Blood pressure | Day 1
  Brachial and central blood pressures
Arterial stiffness | Day 1
  Measured as carotid-femoral pulse wave velocity
Body composition | Day 1
  Whole body and regional lean and fat mass, measure with dual energy X-ray absorptiometry
Cardiorespiratory fitness | Day 1
  Peak oxygen consumption during bicycle ergometry test to volitional fatigue
Blood DNA analysis | Day 1
  Measurement of single-nucleotide polymorphisms associated with NAFLD risk
Liver steatosis | Day 1
  Use of Fibroscan to measure controlled attenuation parameter (measure of steatosis)
Liver fibrosis | Day 1
  Use of Fibroscan to measure elastic modulus (surrogate measure of fibrosis)

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Short, PhD, Principal Investigator — University of Oklahoma
Locations (1):
- University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: Undecided